CLINICAL TRIAL: NCT05017311
Title: Optimized Predictive Treatment In Medications for Unipolar Major Depression (OPTIMUM-D)
Acronym: CAN-BIND-17
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Unity Health Toronto (Other); Centre for Addiction and Mental Health (Other); McMaster University (Other); Queen's University (Other); University of Ottawa (Other); University of British Columbia (Other); University of Calgary (Other); McGill University (Other); Dalhousie University (Other); University of Michigan (Other); Simon Fraser University (Other)
Responsible Party: Principal Investigator, Rudolf Uher, Staff Psychiatrist, Independent Investigator, Professor, Nova Scotia Health Authority
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 1027397
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: major depression; major depressive disorder; MDD; escitalopram; brexpiprazole; neuroimaging; genomics; proteomics; metabolomics
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram; Dexetimide; brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Allocation by Predictive Biomarker Algorithm; Escitalopram + Brexpiprazole (Active Comparator): Patients are randomly assigned to the Allocation by Predictive Biomarker Algorithm group. Based on the outcome result from the personalized predictive biomarker algorithm, patients predicted as non-responders to escitalopram monotherapy will receive open-label escitalopram (10-20 mg/d) and blinded brexpiprazole (0.5-2 mg/d) for the first 8 weeks of the study. For the final 4 weeks of the study, patients will continue to receive both medications but the brexpiprazole will no longer be blinded.
  Interventions: Drug: Escitalopram; Drug: Brexpiprazole
- Allocation by Predictive Biomarker Algorithm; Placebo (Placebo Comparator): Patients are randomly assigned to the Allocation by Predictive Biomarker Algorithm group. Based on the outcome result from the personalized predictive biomarker algorithm, patients predicted to respond to escitalopram monotherapy will receive open-label escitalopram (10-20 mg/d) and blinded placebo for the first 8 weeks of the study. For the final 4 weeks of the study, responders will continue to receive open-label escitalopram without the placebo and non-responders will receive a combination of open-label escitalopram and open-label brexpiprazole.
  Interventions: Drug: Escitalopram
- Random Allocation; Escitalopram + Brexpiprazole (Active Comparator): Patients are randomly assigned to the Random Allocation group and then randomly assigned to receive open-label escitalopram (10-20 mg/d) and blinded brexpiprazole (0.5-2 mg/d) for the first 8 weeks of the study. For the final 4 weeks of the study, patients will continue to receive both medications but the brexpiprazole will no longer be blinded.
  Interventions: Drug: Escitalopram; Drug: Brexpiprazole
- Random Allocation; Placebo (Placebo Comparator): Patients are randomly assigned to the Random Allocation group and then randomly assigned to receive open-label escitalopram (10-20 mg/d) and blinded placebo for the first 8 weeks of the study. For the final 4 weeks of the study, responders will continue to receive open-label escitalopram without the placebo and non-responders will receive a combination of open-label escitalopram and open-label brexpiprazole.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — All patients will receive open-label escitalopram (10-20 mg/d) for the entire study duration (12 weeks).
  Other Names: Cipralex
Drug: Brexpiprazole — Depending on the initial randomization process, patients will either receive blinded brexpiprazole (0.5-2 mg/d) for the entire study duration (12 weeks) or for the last 4 weeks of the study if they received the placebo during the first 8 weeks of the study and were non-responders.
  Other Names: Rexulti
  Arms: Allocation by Predictive Biomarker Algorithm; Escitalopram + Brexpiprazole; Random Allocation; Escitalopram + Brexpiprazole

SUMMARY:
This is a study that will test a predictive biomarker algorithm based on results from a previous study. The goal of this study is to integrate clinical, imaging, EEG, and molecular data across 8 sites to predict treatment outcome for patients experiencing a major depressive episode (MDE).

DETAILED DESCRIPTION:
This is a multi-site, randomized study with two treatment phases: a double-blind primary treatment phase of 8 weeks, and an open-label secondary extension phase of 4 weeks. This study aims to test a predictive biomarker algorithm to select medication treatment for patients with major depressive disorder (MDD) based on results from the recently completed Canadian Biomarker Integration Network in Depression (CAN-BIND)-1 study. This will be accomplished through collection of clinical, neurophysiological, and molecular measures from both MDD patients and healthy controls. This is not a study to evaluate efficacy of medications; medications in this study have been approved by Health Canada and are widely used for the treatment of MDD.

In this study, individuals diagnosed with MDD in a current major depressive episode (MDE) will be randomly assigned to one of the two treatment groups: Personalized Assignment group or Random Assignment group. Patients in the Random Assignment group will randomly receive open-label escitalopram with the addition of either blinded placebo or brexpiprazole for 8 weeks. Patients in the Personalized Assignment group will receive open-label escitalopram with the addition of either placebo or blinded brexpiprazole for 8 weeks depending on what the predictive biomarker algorithm suggests.

At Week 8, participants will be assessed for treatment response (defined as a ≥50% reduction in Montgomery Asberg Depression Rating Scale score). All patients who initially received both open-label escitalopram and blinded brexpiprazole (regardless of treatment group) will continue to receive these medications for another 4 weeks but the brexpiprazole will no longer be blinded. For those patients who initially received open-label escitalopram and blinded placebo (regardless of treatment group), nonresponders will receive open-label escitalopram and open-label brexpiprazole for another 4 weeks and responders will receive open-label escitalopram only for another 4 weeks.

Over the 12 weeks, participants will attend 7 study visits where they will complete clinical assessments (clinician administered and self-report) and cognitive tests; provide blood, urine, and stool samples; undergo neuroimaging procedures (MRI and EEG); and provide speech samples. At the end of the study, modeling methods will be used to integrate data from these measures to determine the features that best predict treatment outcome.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Outpatients 18 to 65 years of age.
* Meet DSM-5 criteria for MDE in MDD as determined by SCID-5.
* Free of psychotropic medications for at least 5 half-lives (e.g. 1 week for most antidepressants, 5 weeks for fluoxetine) before baseline Visit 1 (exceptions: stable use of hypnotics; stable use of stimulants for attention-deficit/hyperactive disorder).
* MADRS score ≥ 24.
* Fluency in English, sufficient to complete the interviews and self-report questionnaires.

Exclusion Criteria:

* Any diagnosis, other than MDD, that is considered the primary diagnosis.
* Bipolar I or Bipolar-II diagnosis.
* Presence of a significant Axis II diagnosis (borderline, antisocial).
* High suicidal risk, defined by clinician judgment.
* Substance dependence/abuse in the past 6 months.
* Presence of significant neurological disorders, head trauma, or other unstable medical conditions.
* Pregnant or breastfeeding.
* Failure of 4 or more adequate pharmacologic interventions (as determined by the Antidepressant Treatment History Form).
* Started psychological treatment within the past 3 months with the intent of continuing treatment.
* Patients who have previously failed escitalopram or showed intolerance to escitalopram or brexpiprazole, and patients at risk for hypomanic switch (i.e. with a history of antidepressant induced hypomania).

Healthy Comparison (HC) Participants

Inclusion Criteria:

* 18 to 65 years of age.
* No history of psychiatric disorders (as determined by SCID-5) or significant physical conditions (e.g. arthritis, fibromyalgia).
* Fluency in English, sufficient to complete the interviews and self-report questionnaires.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Montgomery Asberg Depression Rating Scale (MADRS) scores from baseline | Baseline to Week 8
  Measured as clinical response, defined as a decrease in Montgomery Asberg Depression Rating Scale (MADRS) score at the Week 8 visit, by 50% or greater, from MADRS score at Baseline visit (i.e., lower MADRS scores = better outcome)

SECONDARY OUTCOMES:
Clinical response | Baseline to Week 8
  Defined as a decrease in MADRS score at the Week 8 visit, by 50% or greater, from MADRS score at Baseline visit
Time to clinical response | Baseline to Week 8
  Defined as time (i.e., number of weeks) to achieve clinical response (i.e., decrease in MADRS score at the Week 8 visit, by 50% or greater, from MADRS score at Baseline visit)
Remission at Week 8 | Week 8
  Defined as MADRS score ≤10 at Week 8

OTHER OUTCOMES:
Week 12 clinical outcome - Response | Baseline to Week 8 and Week 8 to Week 12
  Response at Week 12 - defined as a decrease in MADRS score at the Week 12 visit, by 50% or greater, from MADRS score at Baseline visit and Week 8
Week 12 clinical outcome - Remission | Week 12
  Defined as MADRS score ≤10 at Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Uher, MD, Principal Investigator — Nova Scotia Health Authority
Locations (7):
- Canada (7):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University Health Network, Toronto, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
This study is funded by the Ontario Brain Institute (OBI). Data collected from this study is entered into a research database called "Brain-CODE", deployed at a High Performance Computer Virtual Lab (HPCVL). The HPCVL supports the regulatory-compliant (e.g. 21 CRF Part 11, HIPPA, PIPEDA) processes for securing privacy of healthcare data.
Supporting Information: Study Protocol
Time Frame: Within 12 months of study completion.
Access Criteria: By application.
URL: https://braininstitute.ca/research-data-sharing/depression

REFERENCES:
- [Background] Lam RW, Milev R, Rotzinger S, Andreazza AC, Blier P, Brenner C, Daskalakis ZJ, Dharsee M, Downar J, Evans KR, Farzan F, Foster JA, Frey BN, Geraci J, Giacobbe P, Feilotter HE, Hall GB, Harkness KL, Hassel S, Ismail Z, Leri F, Liotti M, MacQueen GM, McAndrews MP, Minuzzi L, Muller DJ, Parikh SV, Placenza FM, Quilty LC, Ravindran AV, Salomons TV, Soares CN, Strother SC, Turecki G, Vaccarino AL, Vila-Rodriguez F, Kennedy SH; CAN-BIND Investigator Team. Discovering biomarkers for antidepressant response: protocol from the Canadian biomarker integration network in depression (CAN-BIND) and clinical characteristics of the first patient cohort. BMC Psychiatry. 2016 Apr 16;16:105. doi: 10.1186/s12888-016-0785-x. PMID 27084692
- [Background] Kennedy SH, Lam RW, Rotzinger S, Milev RV, Blier P, Downar J, Evans KR, Farzan F, Foster JA, Frey BN, Giacobbe P, Hall GB, Harkness KL, Hassel S, Ismail Z, Leri F, McInerney S, MacQueen GM, Minuzzi L, Muller DJ, Parikh SV, Placenza FM, Quilty LC, Ravindran AV, Sassi RB, Soares CN, Strother SC, Turecki G, Vaccarino AL, Vila-Rodriguez F, Yu J, Uher R; CAN-BIND Investigator Team. Symptomatic and Functional Outcomes and Early Prediction of Response to Escitalopram Monotherapy and Sequential Adjunctive Aripiprazole Therapy in Patients With Major Depressive Disorder: A CAN-BIND-1 Report. J Clin Psychiatry. 2019 Feb 5;80(2):18m12202. doi: 10.4088/JCP.18m12202. PMID 30840787
- [Background] Farzan F, Atluri S, Frehlich M, Dhami P, Kleffner K, Price R, Lam RW, Frey BN, Milev R, Ravindran A, McAndrews MP, Wong W, Blumberger D, Daskalakis ZJ, Vila-Rodriguez F, Alonso E, Brenner CA, Liotti M, Dharsee M, Arnott SR, Evans KR, Rotzinger S, Kennedy SH. Standardization of electroencephalography for multi-site, multi-platform and multi-investigator studies: insights from the canadian biomarker integration network in depression. Sci Rep. 2017 Aug 7;7(1):7473. doi: 10.1038/s41598-017-07613-x. PMID 28785082
- [Background] Lopez JP, Fiori LM, Cruceanu C, Lin R, Labonte B, Cates HM, Heller EA, Vialou V, Ku SM, Gerald C, Han MH, Foster J, Frey BN, Soares CN, Muller DJ, Farzan F, Leri F, MacQueen GM, Feilotter H, Tyryshkin K, Evans KR, Giacobbe P, Blier P, Lam RW, Milev R, Parikh SV, Rotzinger S, Strother SC, Lewis CM, Aitchison KJ, Wittenberg GM, Mechawar N, Nestler EJ, Uher R, Kennedy SH, Turecki G. MicroRNAs 146a/b-5 and 425-3p and 24-3p are markers of antidepressant response and regulate MAPK/Wnt-system genes. Nat Commun. 2017 May 22;8:15497. doi: 10.1038/ncomms15497. PMID 28530238
- [Background] Uher R, Frey BN, Quilty LC, Rotzinger S, Blier P, Foster JA, Muller DJ, Ravindran AV, Soares CN, Turecki G, Parikh SV, Milev R, MacQueen G, Lam RW, Kennedy SH; CAN-BIND Investigator Team. Symptom Dimension of Interest-Activity Indicates Need for Aripiprazole Augmentation of Escitalopram in Major Depressive Disorder: A CAN-BIND-1 Report. J Clin Psychiatry. 2020 Jun 16;81(4):20m13229. doi: 10.4088/JCP.20m13229. PMID 32558407
- [Background] Allen TA, Harkness KL, Lam RW, Milev R, Frey BN, Mueller DJ, Uher R, Kennedy SH, Quilty LC. Interactions between neuroticism and stressful life events predict response to pharmacotherapy for major depression: A CAN-BIND 1 report. Personal Ment Health. 2021 Nov;15(4):273-282. doi: 10.1002/pmh.1514. Epub 2021 May 18. PMID 34008342
- [Background] Nogovitsyn N, Muller M, Souza R, Hassel S, Arnott SR, Davis AD, Hall GB, Harris JK, Zamyadi M, Metzak PD, Ismail Z, Downar J, Parikh SV, Soares CN, Addington JM, Milev R, Harkness KL, Frey BN, Lam RW, Strother SC, Rotzinger S, Kennedy SH, MacQueen GM. Hippocampal tail volume as a predictive biomarker of antidepressant treatment outcomes in patients with major depressive disorder: a CAN-BIND report. Neuropsychopharmacology. 2020 Jan;45(2):283-291. doi: 10.1038/s41386-019-0542-1. Epub 2019 Oct 14. PMID 31610545
- [Background] Chakrabarty T, McInerney SJ, Torres IJ, Frey BN, Milev RV, Muller DJ, Rotzinger S, Kennedy SH, Lam RW; CAN-BIND Investigator Team. Cognitive Outcomes with Sequential Escitalopram Monotherapy and Adjunctive Aripiprazole Treatment in Major Depressive Disorder: A Canadian Biomarker Integration Network in Depression (CAN-BIND-1) Report. CNS Drugs. 2021 Mar;35(3):291-304. doi: 10.1007/s40263-021-00793-1. Epub 2021 Mar 8. PMID 33683582
- [Background] Morton E, Bhat V, Giacobbe P, Lou W, Michalak EE, McInerney S, Chakrabarty T, Frey BN, Milev RV, Muller DJ, Parikh SV, Rotzinger S, Kennedy SH, Lam RW; CAN-BIND Investigator Team. Predictors of Quality of Life Improvement with Escitalopram and Adjunctive Aripiprazole in Patients with Major Depressive Disorder: A CAN-BIND Study Report. CNS Drugs. 2021 Apr;35(4):439-450. doi: 10.1007/s40263-021-00803-2. Epub 2021 Apr 16. PMID 33860922
- [Background] Ayyash S, Davis AD, Alders GL, MacQueen G, Strother SC, Hassel S, Zamyadi M, Arnott SR, Harris JK, Lam RW, Milev R, Muller DJ, Kennedy SH, Rotzinger S, Frey BN, Minuzzi L, Hall GB; CAN-BIND Investigator Team. Exploring brain connectivity changes in major depressive disorder using functional-structural data fusion: A CAN-BIND-1 study. Hum Brain Mapp. 2021 Oct 15;42(15):4940-4957. doi: 10.1002/hbm.25590. Epub 2021 Jul 23. PMID 34296501
- [Background] Caspani G, Turecki G, Lam RW, Milev RV, Frey BN, MacQueen GM, Muller DJ, Rotzinger S, Kennedy SH, Foster JA, Swann JR. Metabolomic signatures associated with depression and predictors of antidepressant response in humans: A CAN-BIND-1 report. Commun Biol. 2021 Jul 22;4(1):903. doi: 10.1038/s42003-021-02421-6. PMID 34294869
- [Background] Allen TA, Lam RW, Milev R, Rizvi SJ, Frey BN, MacQueen GM, Muller DJ, Uher R, Kennedy SH, Quilty LC. Early change in reward and punishment sensitivity as a predictor of response to antidepressant treatment for major depressive disorder: a CAN-BIND-1 report. Psychol Med. 2019 Jul;49(10):1629-1638. doi: 10.1017/S0033291718002441. Epub 2018 Sep 17. PMID 30220263
- [Background] Alders GL, Davis AD, MacQueen G, Strother SC, Hassel S, Zamyadi M, Sharma GB, Arnott SR, Downar J, Harris JK, Lam RW, Milev R, Muller DJ, Ravindran A, Kennedy SH, Frey BN, Minuzzi L, Hall GB; CAN-BIND Investigator Team. Escitalopram ameliorates differences in neural activity between healthy comparison and major depressive disorder groups on an fMRI Emotional conflict task: A CAN-BIND-1 study. J Affect Disord. 2020 Mar 1;264:414-424. doi: 10.1016/j.jad.2019.11.068. Epub 2019 Nov 13. PMID 31757619
- [Background] Chakrabarty T, Harkness KL, McInerney SJ, Quilty LC, Milev RV, Kennedy SH, Frey BN, MacQueen GM, Muller DJ, Rotzinger S, Uher R, Lam RW. Childhood maltreatment and cognitive functioning in patients with major depressive disorder: a CAN-BIND-1 report. Psychol Med. 2020 Nov;50(15):2536-2547. doi: 10.1017/S003329171900268X. Epub 2019 Oct 4. PMID 31583989
- [Background] Dunlop K, Rizvi SJ, Kennedy SH, Hassel S, Strother SC, Harris JK, Zamyadi M, Arnott SR, Davis AD, Mansouri F, Schulze L, Ceniti AK, Lam RW, Milev R, Rotzinger S, Foster JA, Frey BN, Parikh SV, Soares CN, Uher R, Turecki G, MacQueen GM, Downar J. Clinical, behavioral, and neural measures of reward processing correlate with escitalopram response in depression: a Canadian Biomarker Integration Network in Depression (CAN-BIND-1) Report. Neuropsychopharmacology. 2020 Jul;45(8):1390-1397. doi: 10.1038/s41386-020-0688-x. PMID 32349119
- [Background] Yrondi A, Fiori LM, Frey BN, Lam RW, MacQueen GM, Milev R, Muller DJ, Foster JA, Kennedy SH, Turecki G. Association Between Side Effects and Blood microRNA Expression Levels and Their Targeted Pathways in Patients With Major Depressive Disorder Treated by a Selective Serotonin Reuptake Inhibitor, Escitalopram: A CAN-BIND-1 Report. Int J Neuropsychopharmacol. 2020 Feb 1;23(2):88-95. doi: 10.1093/ijnp/pyz066. PMID 31819986
- [Background] McInerney SJ, Chakrabarty T, Maciukiewicz M, Frey BN, MacQueen GM, Milev RV, Ravindran AV, Rotzinger S, Kennedy SH, Lam RW; CAN-BIND Investigator Team. Cognition and Its Association with Psychosocial and Occupational Functioning during Treatment with Escitalopram in Patients with Major Depressive Disorder: A CAN-BIND-1 Report: La Cognition Et Son Association Avec Le Fonctionnement Psychosocial Et Professionnel Durant Le Traitement Par Escitalopram Chez Des Patients Souffrant De Trouble Depressif Majeur: Une Etude Can-Bind-1. Can J Psychiatry. 2021 Sep;66(9):798-806. doi: 10.1177/0706743720974823. Epub 2020 Dec 23. PMID 33353384